CLINICAL TRIAL: NCT07053059
Title: Phase 2 Study Assessing the Clinical Activity and Safety of Obecabtagene Autoleucel as a Consolidation in Patients With Newly Diagnosed High-risk B-cell Acute Lymphocytic Leukemia (ALL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Autolus, Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0580; NCI-2025-04660 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphocytic Leukemia (ALL)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Obecabtagene Autoleucel (Experimental): Participants in morphological remission will be eligible in the present study, the dose of obe-cel will be as per the FELIX trial as follows:
  Interventions: Drug: Obecabtagene autoleucel

INTERVENTIONS:
Drug: Obecabtagene autoleucel — given by Infusion

SUMMARY:
The goal of this clinical research study is to learn if obecabtagene autoleucel (obe-cel) can help to control newly diagnosed, high-risk B-cell ALL when given as consolidation therapy. Consolidation therapy is given after the first phase of treatment.

DETAILED DESCRIPTION:
Primary Objectives To assess the Efficacy of Obecabtagene autoleucel [anti-CD19 autologous derived chimeric antigen receptor T-cell (CAR-T)] in terms of EFS in patients with newly diagnosed high-risk B-cell ALL (defined by baseline high-risk genomics or persistent MRD) post cytoreductive chemoimmunotherapy: 18-month EFS

Secondary Objectives:

1. 24-month overall survival (OS)
2. For Ph-negative B-cell ALL: Rate of persistent MRD negativity by flow cytometry and NGS at 18 months
3. For Ph-positive B-cell ALL: Rate of persistent MRD negativity by flow cytometry, NGS and BCR::ABL1 qPCR (CMR) at 18 months
4. Achievement of BCR::ABL1 complete molecular response (CMR) in patients with Ph-positive ALL having persistent measurable disease at any level before obe-cel infusion
5. Achievement of NGS MRD negativity amongst patients in CR and not MRD negative before obe-cel
6. Time to initiation of next anti-leukemia therapy except HSCT when done in ongoing continued morphological response (patients who did not start next anti-leukemia therapy except HSCT will be censored at the last follow-up/death).
7. Rates of HSCT in morphologic remission after obe-cel infusion
8. Safety

Exploratory Objectives:

1. CAR-T-cell expansion by digital droplet PCR (ddPCR) assay by a manufacturer designated central laboratory (CellCarta) on Days 7, 14, 21, 28, 3 months and then every 3 months up to 12 months post infusion. This will be a send-out test.
2. B-cell aplasia (Days 0, 7, 14, 28, monthly up to 3 months and then every 3 months up to 24 months post infusion)
3. Measurable residual disease (MRD) negativity by next-generation sequencing (NGS) (at 1 in 105-6 sensitivity) (PB on D14 and PB/BM: Day 28, and then Q3 months up to 24 months post infusion)
4. Cytokine panel to study cytokine profile including IL1, IL6, IFNG, TNFalpha from infusion (Days 0, 1, 2, 4, 7, 10, 14, 28)
5. Additional correlatives samples to address tumor samples and immune system factors will be collected at baseline, D28 and Q3 months from infusion. These include samples for bulk RNA sequencing of the tumor and germline and single cell RNA sequencing of CAR T-cells as also for assessing the methylation signatures of the CAR T-cells.

risk B-cell ALL (defined by baseline high-risk genomics or persistent MRD) post cytoreductive chemoimmunotherapy: 18-month EFS

ELIGIBILITY:
Inclusion Criteria:

I. Patients of age .18 years with high-risk B-cell ALL in first remission and <5% BM blasts with at least one high-risk feature defined as:

a. Ph-negative B-cell ALL: i. KMT2A rearranged ALL ii. Complex cytogenetics as per NCCN 2022 iii. Low-hypodiploidy/tetraploidy iv. Philadelphia-like ALL (based on CRLF2 overexpression or recurrent Ph-like genetic fusions) v. TP53 mutation (variant allele fraction >2%) vi. Persistent MRD by flow cytometry and/or NGS b. Ph-positive B-cell ALL: i. IKZF1plus genotype (IKZF1 deletion coexisting with PAX5 or CDKN2A/2B, or PAR1 region deletions) or other high-risk features such as VPRB1 deletion, etc. ii. High WBC (>30 x 109/L) at initial presentation iii. Persistent MRD by flow cytometry and/or NGS and/or PCR II. Performance status of 0, 1, or 2 III. Adequate organ function with creatinine less than or equal to 1.6 mg/dl, bilirubin less than or equal to 3.5 mg and ALT and AST less than or equal to 5 times institutional upper limit of normal IV. Patients should be CD19 expression positive (>1%) before enrollment VII. Patients with controlled CNS and/or other extramedullary leukemia will be eligible.

Exclusion Criteria:

Pregnant or lactating; women of child-bearing potential (WOCBP) must have negative pregnancy test. WOCBP defined as not post-menopausal for 12 months or no previous surgical sterilization.

Patients with history of Hepatitis B, Hepatitis C, Human Immunodeficiency Virus (HIV) infections, even if under control. (Patients with Hepatitis B core antibody positive alone will not be an exclusion factor if HBV DNA PCR is negative).

Active and uncontrolled disease/infection as judged by the treating physician

Unable or unwilling to sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org